CLINICAL TRIAL: NCT02233257
Title: Expanded Access for Lorenzo's Oil (GTO/GTE) in Adrenoleukodystrophy
Status: No longer available | Type: Expanded Access
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1401M47561
Record Dates: First submitted 2014-05-05; First posted 2014-09-08 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: X-linked Adrenoleukodystrophy
Keywords: Adrenoleukodystrophy; Lorenzo's oil; erucic acid
MeSH Terms: conditions — Adrenoleukodystrophy | interventions — Lorenzo's oil; trierucate

INTERVENTIONS:
Drug: Lorenzo's Oil — Oral use of Lorenzo's oil to lower very long chain fatty acids
  Other Names: Glyceryl trierucate

SUMMARY:
X-linked adrenoleukodystrophy (ALD) is a genetic disorder affecting the brain and adrenal glands. Approximately one third of boys who are at risk will develop cerebral disease. Using a specific diet and the compound Lorenzo's oil, it can be shown that very long chain fatty acids may be lowered in the blood, but it is not known to what degree that may prevent the onset of childhood disease.

This proposal makes available Lorenzo's oil to individuals with ALD, a life threatening disorder for which there are presently no other therapies.

DETAILED DESCRIPTION:
Expanded Access for Lorenzo's Oil in X-linked Adrenoleukodystrophy to Intermediate Size Group

Introduction/Rationale: A diet that consists predominantly of long-chain monounsaturated fatty acids has been demonstrated to reduce the levels of very long chain fatty acids (VLCA) in individuals with X-linked adrenoleukodystrophy (ALD). VLCFA are the primary biochemical abnormality in this genetic disorder and have been implicated in the pathogenesis of the cerebral disease. It has been demonstrated in an open study that reduction of VLCFA for more than a year is protective for childhood cerebral disease.

The purpose of this expanded access proposal is to transition an open label study presently ongoing in boys between the ages of 18 months and 13 years of age to an expanded access study. The reason for this transition is lack of funding for the investigator to continue to support this as a study. A study requires investigator involvement including the assistance of research associates to monitor and track outcomes, perform neuropsychological assessments, monitor adverse events, and coordinate periodic evaluations.

A move to expanded access would decentralize the coordination and monitoring of evaluations which are clinically indicated even for participants who are not participating in a study. This role would be undertaken by the treating physician.

Data collected in such an open study could serve as safety material for a later filing.

Study Population:

* Males with X-linked adrenoleukodystrophy; see inclusion/exclusion criteria below.

Procedure:

1. Individuals who wish to obtain oil will submit clinical documentation of diagnosis to Dr. Gerald Raymond. This will be either elevated very long chain fatty acids (VLCFA) or DNA diagnosis of a mutation.
2. Identify a provider who will be responsible for the supervision of the diet. It is suggested that this be an individual who is experienced in managing individuals on a special diets such as a biochemical geneticist or neurologist with experience in ALD.
3. Studies required before prescription (It is important to emphasize that while many of the following are performed solely for the use of Lorenzo's oil, the costs of these investigations and consults will be the financial responsibility of the participants.)

   1. Baseline VLCFA, complete blood count with platelets, and comprehensive metabolic panel
   2. Nutrition consult with a determination of daily calories. Thirty percent of calories will be provided by lipids and 2/3 of these lipid calories will be provided by long chain monounsaturated fatty acids (Lorenzo's oil). This nutritional evaluation will include the following.

   i. Present body parameters including weight, height, and BMI ii. Calculated daily calories and other nutritional needs for growth. iii. Calculation of percent of diet as lipids and amount of oil to be consumed daily iv. Instruction in diet restriction and monitoring of said diet. v. Recommend supplements. vi. Instructions in providing diet recall vii. Suggestions for maintaining and improving compliance. c. An MRI and adrenal testing are clinically indicated and will be required as part of expanded access.
4. Clinical research forms (CRF) will be designed for the baseline and follow up information for uniformity of documentation.
5. Upon receipt of this information, Dr. Raymond will provide an authorization of the prescription to the supplier, Nutricia N.A.
6. Monitoring while receiving oil will consist of the following

   1. VLCFA; Complete blood count (CBC), and Comprehensive metabolic panel every 3 months
   2. Nutrition consult yearly.
   3. Magnetic Resonance Imaging of the brain will be performed every 6-12 months
   4. Appropriate monitoring of adrenal function.
   5. CRFs' will be forwarded every three months for all active participants on a January, April, July, October schedule
   6. The identified provider will be responsible for providing this information to Dr. Raymond's office. Failure to provide this information will result in withholding of authorization and no dispensing of the product.
   7. No more than 3 months' supply of the product will be authorized or shipped at a time.
   8. In the event of development of thrombocytopenia, Lorenzo's oil will be suspended and glyceryl trioleate (GTO) substituted for one month and then reintroduced as half dose of Lorenzo's oil followed by incremental increases as tolerated. We have previously used 80,000 platelets as a lower limit and would recommend this as providing an adequate margin of safety.
7. Adverse events will be tracked and if resulting in hospitalization or death will be reported as required to the sponsor and FDA in the required period of time.

Otherwise all reported adverse events will be tabulated and reported in the yearly IND report.

Adverse events will include conversion of normal MRIs to those demonstrating cerebral disease and any interventions including bone marrow transplantation or gene therapy which are presently the only options to halt cerebral disease.

ELIGIBILITY:
Inclusion Criteria:

* Males with X-linked adrenoleukodystrophy as determined by biochemical or genetic determination.
* Greater than 18 months of age through 18 years of age
* Normal cerebral MRI at baseline.

Exclusion Criteria:

* Medical issues which preclude the administration of Lorenzo's oil

Ages: 18 Months to 18 Years | Sex: Male
Age Groups: Child, Adult

CONTACTS AND LOCATIONS:
Overall Officials: Gerald V Raymond, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Medical Center, Minneapolis, Minnesota, United States